CLINICAL TRIAL: NCT04494568
Title: Evaluation of High Intensity Focused Ultrasound (HIFU) in the Treatment of Rectal Endometriosis
Acronym: ENDO-HIFU-R1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EDAP TMS S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU-F-20.01
Record Dates: First submitted 2020-07-22; First posted 2020-07-31 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Endometriosis, Rectum
Keywords: rectal endometriosis, HIFU
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: INTERVENTIONAL, PROSPECTIVE, MULTICENTRIC, NON-RANDOMIZED AND NON-CONROLLED STUDY
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIFU intervention (Experimental): patients will benefit of an HIFU Treatment of their rectal endometriosis
  Interventions: Device: HIFU treatment

INTERVENTIONS:
Device: HIFU treatment — HIFU Treatment of rectal endometriosis

SUMMARY:
Rectal endometriosis (RE) induces lesions associated with painful symptoms that can alter quality of life. High Intensity Focused Ultrasound (HIFU) is a non-invasive ablative procedure using a high-intensity ultrasound probe to induce tissue devitalization using acoustic cavitation and thermal ablation. Focal One® is a transrectal HIFU device, which is validated to treat prostatic cancer.

The primary objective of this clinical investigation is to evaluate the safety of the HIFU treatment of rectal endometriosis with Focal One® HIFU device.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged at least 25 years-old
* Rectal endometriosis in preoperative imaging, without other digestive locations (colon, ileum and small intentine)
* Symptomatic patient refusing hormonal treatment and/or surgery.
* Endometriosic nodule visible on echography with contrast and confirmed in Gadolinium MRI and difusion sequence (according to standardized protocol)
* Nodule with intrarectal protrusion of less than 50% (allowing the positioning of the probe in front of the rectal nodule)
* Distance from the upper pole to the anal margin ≤ 15 cm (measurement by MRI with intra-rectal contrast)
* No curent pregnancy (negative BHCG <72h before the HIFU procedure) and no pregnancy project within 6 months after the HIFU procedure (post-treatment MRI delay)
* Patient agreeing not to change her hormone treatment for the duration of the study.
* Patient accepting the study constraints
* Health insurance affiliated patient or beneficiary of an equivalent coverage

Exclusion Criteria:

* Virgin patient
* Ongoing uro-genital infection
* Anorectal anatomy incompatible with HIFU therapy
* History of segmental rectal resection with mechanical anastomosis, shaving or discoid resection
* Patient with an implant within 1cm of the treatment area (stent, catheter, ESSURE® contraceptive implants).
* Inflammatory colon disease (ulcerative colitis, Crohn's disease and others)
* Latex allergy
* Patient with contraindications to MRI
* Patient with contraindications to Gadolinium injection
* Patient previously treated with HIFU for a rectal endometriotic lesion
* Patient not speaking nor reading French
* Patient deprived of liberty following a legal or administrative decision
* Patient under guardianship or tutelage measure

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the tolerance of rectal endometriosis treatment with HIFU | 6 months
  The tolerance of the treatment will be evaluated by the analysis of adverse events occurrence at 6 months post-HIFU treatment

SECONDARY OUTCOMES:
Evaluation of the gynecological symptoms evolution of patients after HIFU treatment | at 1 month, 3 months and 6 months post-intervention
  EVA symptom Questionnaires
Evaluation of the of quality of life evolution of patients after HIFU treatment | at 1 month, 3 months and 6 months post-intervention,
  Quality of life questionnaire : MOS- SF-36
Evaluation of the evolution of the nodule's volume | at 6 months
  The pre- and post-treatment comparison of the volume of the endometriodsis nodule measurement.
Evaluation of the post-intervention analgesic treatment | during the fisrt 10 days post treatment.
  The level of medication during the fisrt 10 days post treatment will be studied by analysing the data collected in patient book.
Evaluation of the digestive symptoms evolution of patients after HIFU treatment | at 1 month, 3 months and 6 months post-intervention
  Wexner
Evaluation of the digestive symptoms evolution of patients after HIFU treatment | at 1 month, 3 months and 6 months post-intervention
  Kess questionnaires
Evaluation of the sexual symptoms evolution of patients after HIFU treatment | at 1 month, 3 months and 6 months post-intervention
  SFSI questionnaire
Evaluation of the urinary symptoms evolution of patients after HIFU treatment | at 1 month, 3 months and 6 months post-intervention
  USP questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gil DUBERNARD, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (5):
- France (5):
  - CHU de Angers, Angers
  - Clinique Tivoli-Ducos, Bordeaux
  - Hôpital BICETRE, Le Kremlin-Bicêtre
  - Clinique de Gynécologie, Lille
  - Hopital de la Croix Rousse, Lyon

REFERENCES:
- [Derived] Dubernard G, Maissiat E, Legendre G, Dennis T, Capmas P, Warembourg S, Descamps P, Chavrier F, Roman H, Fernandez H, Nguyen-Ba E, Merlot B, Rousset P, Lafon C, Philip CA. Evaluating the safety of high-intensity focused ultrasound treatment for rectal endometriosis: results from a French prospective multicentre study including 60 patients. Hum Reprod. 2024 Aug 1;39(8):1673-1683. doi: 10.1093/humrep/deae127. PMID 38914481